CLINICAL TRIAL: NCT00924157
Title: Effect of a Protein Hydrolysate Rich in Lacto-tripeptide (IPP) on Hyperemic Blood Flow and Flow-mediated Dilation in Patients With Coronary Artery Disease
Brief Title: Effect of Ile-Pro-Pro (IPP) on Endothelial Function in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Joseph A. Vita, Professor of Medicine, Boston University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-27820
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — indolepropanol phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: IPP — Protein hydrolysate rich in lacto-tripeptide (IPP) up to 5 to 15 mg/day
Other: Placebo — Matching placebo capsules

SUMMARY:
This study will investigate whether the lacto-tripeptide Ile-Pro-Pro (IPP) improves the function of the endothelium in patients with coronary artery disease. The study has a crossover design. Participants will be treated with a protein hydrolysate rich in IPP for 12 weeks and placebo for 12 weeks with a four-week rest period between treatment periods. The investigators will use ultrasound to test the function of the endothelium in the brachial artery before, after 6 weeks, and after 12 weeks of each treatment. Blood will be collected before and after each treatment. The investigators hypothesize that IPP will improve endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease

Exclusion Criteria:

* Treatment with an ACE inhibitor or ARB
* Pregnancy
* Other major illness
* Treatment with an investigational drug within 4 weeks

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Brachial Artery Flow-Mediated Dilation and Reactive Hyperemia | 12 weeks

SECONDARY OUTCOMES:
Carotid-Femoral Pulse Wave Velocity | 12 weeks
Leg Reactive Hyperemia | 12 weeks
Digital Pulse Amplitude Tonometry | 12 weeks
Blood pressure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Vita, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States